CLINICAL TRIAL: NCT04497792
Title: A Long-term, Randomized Study to Evaluate the Effects of Empagliflozin in Combination With Standard Hypoglycemic Therapy on Early and Long-term Results of Planned Percutaneous Coronary Interventions in Patients With Type 2 Diabetes.
Brief Title: Safety and Efficacy of Empagliflozin for Patients With Diabetes Mellitus and Planned Percutaneous Coronary Interventions
Acronym: SAFARY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Responsible Party: Principal Investigator, Olga Barbarash, Principal, Research Institute for Complex Problems of Cardiovascular Diseases, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16_001
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus; Percutaneous Coronary Intervention
Keywords: stable coronary artery disease; empagliflozin
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus | interventions — empagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The treatment group are patients with stable coronary artery disease before planned percutaneous coronary intervention. All of them will receive empagliflozin additionally to previously taken hypoglycemic treatment.
  Interventions: Drug: Empagliflozin 10Mg Tab
- Control group (Other): patients continue previously prescribed medication intake
  Interventions: Drug: hypoglycemic therapy

INTERVENTIONS:
Drug: Empagliflozin 10Mg Tab — Patients from treatment group received empagliflozin 10 mg daily additionally to previously prescribed diabetes medication
  Other Names: metformin
  Arms: Treatment group
Drug: hypoglycemic therapy — hypoglycemic therapy.
  Other Names: metformin
  Arms: Control group

SUMMARY:
Aim: To study the effectiveness and safety of empagliflozin as a preoperative preparation tool, as well as to improve the long-term prognosis of planned percutaneous coronary interventions in patients with type 2 diabetes

DETAILED DESCRIPTION:
Patients with type 2 diabetes will be randomized into 2 groups using the envelope method. One group will receive empagliflozin 10 mg 1 month before planned percutaneous coronary interventions and for 12 months thereafter in addition to previously taken hypoglycemic therapy. Patients of the second group will continue to take previously prescribed hypoglycemic therapy.

Thus, the safety and effectiveness of empagliflozin for preoperative preparation of patients with type 2 diabetes before planned percutaneous coronary interventions will be evaluated, as well as the impact on the immediate and long-term outcomes of percutaneous coronary interventions in comparison with patients on standard hypoglycemic therapy

ELIGIBILITY:
Inclusion Criteria:

* signed inform concent
* stable coronary artery disease
* planned percutaneous coronary intervention
* diabetes mellitus

Exclusion Criteria:

* previously performed coronary revascularization
* glomerular filtration rate less than 45 ml/min
* intolerance to empagliflozin
* serum potassium more than 5/5 mmol/l
* heart failure (NYHA III-IV)
* congenital heart disease
* acute coronary syndrome less than 3 months before enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
glomerular filtration rate(GFR) | baseline-24 weeks
  The glomerular filtration rate(GFR) will be measured at each visit. GFR more than 60 will be recognized as normal.
HbA1C level | baseline-24 weeks
  The HbA1C will be measured (in %) at each visit. HbA1C less than 6.1% will be recognized as normal.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Barbarash, Principal Investigator — Research Institute for complex issues of cardiovascular diseases

IPD SHARING:
Plan to Share IPD: No